CLINICAL TRIAL: NCT04662073
Title: COVID-19 Outpatient Pragmatic Platform Study (COPPS): A Pragmatic Multi-arm, Adaptive, Phase 2, Blinded, Randomized Placebo-controlled Platform Trial to Assess the Efficacy of Different Investigational Therapeutics in Reducing Time to Disease Resolution or Viral Load Cessation, as Compared to Standard Supportive Care in Outpatients With COVID-19
Brief Title: COVID-19 Outpatient Pragmatic Platform Study (COPPS) - Camostat Sub-Protocol
Acronym: COPPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment into the camostat subprotocol was halted prematurely as a result of loss of equipoise due to external findings including those related to monoclonal antibodies.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPPS-Camostat
Record Dates: First submitted 2020-12-08; First posted 2020-12-10 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Outpatient
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Camostat (Experimental): Participants are randomized to receive camostat for 10 days.
  Interventions: Drug: Camostat
- Matching Placebo (Placebo Comparator): Participants are randomized to receive placebo to match camostat for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Camostat — 200 mg (2 x 100 mg tablet) administered orally four times daily (800 mg total daily dose).
  Arms: Camostat
Drug: Placebo — Placebo to match camostat administered orally four times daily
  Arms: Matching Placebo

SUMMARY:
The overall objective of this study is to efficiently evaluate the clinical efficacy and safety of different investigational therapeutics among adults who have COVID-19 but are not yet sick enough to require hospitalization. The overall hypothesis is that through an adaptive trial design, potential effective therapies (single and combination) may be identified for this group of patients.

COVID-19 Outpatient Pragmatic Platform Study (COPPS) is a pragmatic platform protocol designed to evaluate COVID-19 treatments by assessing their ability to reduce viral shedding (Viral Domain) or improve clinical outcomes (Clinical Domain). To be included into the platform, every investigational product will collect data for both Domain primary endpoints. Individual treatments to be evaluated in the platform will be described in separate sub-protocols.

DETAILED DESCRIPTION:
The platform study allows investigational products with objectives either: evaluating viral shedding (Virology Domain); and COVID-19 related Clinical Outcomes (Clinical Domain).

The primary objective for investigational products within the Viral Domain is:

A. To evaluate the efficacy of each therapeutic intervention in addition to standard supportive care (SSC) compared with SSC in reducing viral shedding of SARS-CoV-2 virus in outpatients with COVID-19 disease.

The primary objective for investigational products within for the Clinical Domain is:

B. To evaluate the efficacy of each therapeutic intervention in addition to SSC as compared to SSC in improving sustained clinical outcomes in outpatients with COVID-19 disease.

Secondary objectives are:

1. The objective of the non-assigned domain an investigational product is under.

   1. If under Clinical Domain, reduction in viral shedding.
   2. If under Viral Domain, time to resolution of symptoms.
2. To evaluate the efficacy of each therapeutic intervention in reducing SARS-CoV-2 related hospitalizations, ED visits, or death in outpatients with COVID-19 disease.
3. To assess the development of antibodies against SARS-CoV-2
4. To evaluate the safety and tolerability of each therapeutic intervention compared with placebo (supportive care).

ELIGIBILITY:
Inclusion Criteria:

1. 1. Outpatient setting
2. Age ≥ 18 years and ≤ 80 years at the time of the assessment
3. Able and willing to understand the study, adhere to all study procedures, and provide written informed consent
4. Initial diagnosis of COVID-19 disease as defined by an FDA-cleared molecular diagnostic assay positive for SARS-CoV-2 with no more than 72 hours from the initial swab used in the diagnosis to the time of commencing informed consent.
5. At baseline, at least two symptoms should have mild or higher severity score, where at least one of the mild symptoms is not cough, fatigue, or loss of smell/taste OR at least one symptom has a moderate or higher severity score on the COVID Outpatient Symptom Scale (COSS).
6. Participant's COVID-19 related symptom onset occurred within 7 days prior to time of randomization.
7. Other inclusion criteria specific to the investigational product that may, in the eyes of the investigator, be deemed necessary.

Additional inclusion criteria for camostat protocol:

1. If male, must be sterile, OR agree not to donate semen AND agree to strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
2. If female, must be unable to bear children, OR ensure that their male partner is incapable of fathering a child, OR, if of childbearing potential will strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication, and must agree to stop breast-feeding prior to first dose of study drug and through seven days after completing therapy.

Exclusion Criteria:

1. At screening, the participant needs to be admitted to the hospital or is being evaluated for potential admission.
2. Previous use of experimental drugs that may be active against COVID-19 in the eyes of the investigators.
3. Participant yields a positive urine pregnancy test at screening.
4. Participant is using adrenocorticosteroids (except topical or inhaled preparations or oral preparations equivalent to or less than 10 mg of oral prednisone) or immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers).

   NOTE: Treatment of study participants following institutional COVID-19 treatment policies or guidelines, including the use of immunomodulatory medications, is permitted. This excludes treatment with agents that have the potential for direct antiviral activity, including convalescent plasma and NO, and co-enrollment into other clinical studies that evaluate investigational agents for COVID-19.
5. Participant has a serious chronic disease (e.g., uncontrolled human immunodeficiency virus [HIV], cancer requiring chemotherapy within the preceding 6 months, and/or moderate or severe hepatic insufficiency).
6. Has renal insufficiency including severe renal impairment and ESRD and/or requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD).
7. Has liver impairment greater than Child Pugh A.
8. Has a history of alcohol or drug abuse in the previous 6 months.
9. Has a psychiatric disease that is not well controlled where controlled is defined as: stable on a regimen for more than one year.
10. Has taken another investigational drug within the past 30 days.
11. Is deemed by the Investigator to be ineligible for any reason.

Additional exclusion criteria for camostat protocol:

1. Participant has a history of gout and coagulation disorders.
2. Participant has a concomitant bacterial respiratory infection as documented by a respiratory culture with microbiologic growth. NOTE: Participants on empirical antibiotic treatment for possible but unproven bacterial pneumonia, but who are positive for SARS-CoV-2, are allowed in the study.
3. Has previously received camostat mesilate within the past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Parsonnet, MD, Principal Investigator — Stanford University; Chaitan Khosla, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - ValleyCare Medical Center, Pleasanton, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bunning B, Hedlin H, Purington N, Sundaram V, Kapphahn K, Weng Y, Cunanan K, Maldonado Y, Singh U, Khosla C, O'Hara R, Nicolls M, Springman E, Parsonnet J, Rogers A, Levitt J, Desai M. The COVID-19 Outpatient Pragmatic Platform Study (COPPS): Study design of a multi-center pragmatic platform trial. Contemp Clin Trials. 2021 Sep;108:106509. doi: 10.1016/j.cct.2021.106509. Epub 2021 Jul 16. PMID 34274494

RESULTS

PARTICIPANT FLOW:
Groups:
- Camostat: Participants receive camostat 200 mg (2 x 100 mg tablet) orally four times daily for 10 days.
- Matching Placebo: Participants receive placebo to match camostat for 10 days.
Period: Overall Study
Arm/Group | Camostat | Matching Placebo
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat | Matching Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: For the Viral Domain: Change in Viral Shedding
Description: The number of participants who had viral shedding at Day 10 is reported. Change in shedding of SARS-CoV-2 virus through day 10 attained from self-collected nasal swab RT-PCR data after transformation using a referenced standard curve.
Time Frame: 10 days
Population: No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
Participants | 1 |

2. Secondary Outcome: For Clinical Domain: Time-to-sustained-resolution
Description: The number of participants with sustained resolution by Day 28 is reported. Resolution is defined as the first day where no symptoms are self-reported on all succeeding days through and including day 28, not including sense of taste or smell, and defining recovery for fatigue and cough as mild or none.
Time Frame: 28 days
Population: No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
Participants | 2 |

3. Secondary Outcome: Time to Viral Cessation
Description: Defined as the time in days from randomization to the first of two consecutive negative RT-PCR results of self-collected nasal swabs.
Time Frame: 28 days
Population: No participants were enrolled in the placebo arm..
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
days | NA [NA to NA] — Not calculable due to insufficient number of events |

4. Secondary Outcome: Time to First Resolution
Description: The number of participants with first resolution by Day 28 is reported. First resolution is defined as the first study day where no symptoms are self-reported, not including sense of taste or smell, and defining recovery for fatigue and cough as mild or none.
Time Frame: 28 days
Population: No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
Participants | 2 |

5. Secondary Outcome: Time to Full Resolution
Description: The number of participants with full resolution by Day 28 is reported. Full resolution is defined as the study day where no symptoms are first self-reported.
Time Frame: 28 days
Population: No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
Participants | 2 |

6. Secondary Outcome: Indicator of SARS-CoV-2 Related Hospitalizations, ED Visits, or Death in Outpatients With COVID-19 Disease.
Description: Count (%) of participants that experienced SARS-CoV-2 a related hospitalization, emergency department (ED) visit, or death.
Time Frame: 28 days
Population: No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

7. Secondary Outcome: Indicator Participant Has Developed Antibodies to SARS-CoV-2
Time Frame: 28 days
Population: No antibody results data were collected in the camostat arm, and no participants were enrolled in the placebo arm.
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Indicator Participant Has a Negative SARS-CoV2 RT-PCR Test
Description: Count (%) of participants with a negative SARS-CoV2 RT-PCR test at day 14
Time Frame: day 14
Population: Participants with data collected. No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 |

9. Secondary Outcome: Indicator Participant Has a Negative SARS-CoV2 RT-PCR Test
Description: Count (%) of participants with a negative SARS-CoV2 RT-PCR test at day 28
Time Frame: day 28
Population: Participants with data collected. No participants were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Matching Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 |

ADVERSE EVENTS:
Time Frame: 10 months
Description: Safety Analysis Set: per protocol, the safety analysis was performed using the as-treated population and includes all patients who received study treatment. As pre-specified in the study protocol, any clinical events related to the progression of COVID-19 (except death) would not be considered adverse events.
Arm/Group | Camostat | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment and did not achieve statistical power as specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Master Protocol, Amendent 7 (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT04662073/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Camostat Sub-Study, Amendment 4 (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT04662073/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Master Protocol, Amendent 9 (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04662073/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Camostat Sub-Study, Amendment 6 (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04662073/Prot_SAP_003.pdf